CLINICAL TRIAL: NCT00085163
Title: Multicenter, Double-Blind, Placebo-Controlled Randomized Phase III Study of Adjuvant Therapy With Celecoxib in Combination With Chemotherapy in Patients With Curatively Resected Stage III Colon Cancer
Brief Title: Celecoxib Combined With Fluorouracil and Leucovorin in Treating Patients With Resected Stage III Adenocarcinoma (Cancer) of the Colon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Dutch Colorectal Cancer Group (DCCG) (Unknown); Arbeitsgemeinschaft fur Internistische Onkologie (Other); Onkologie (Unknown); Egyptian Foundation For Cancer Research (Other); EORTC GI Group (EORTC 40023) (Unknown); Federation Francophone de Cancerologie Digestive (Other); GCCD-APIO - Grupo Cooperativo do Cancro Digestivo da Associação Portuguesa de Investigação (Unknown); Oncológica (Unknown); Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other); GOCCI - Gruppo Oncologico Chirurgico Cooperativo Italiano (Unknown); GOIRC - Gruppo Oncologico Italiano di Ricerca Clinica (Unknown); SG - Scandinavian Group (Unknown); TTD - Grupo Español para el Tratamiento de Tumores Digestivos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: EORTC-40023; EORTC-40023; PETACC-5
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Celecoxib; Fluorouracil; Leucovorin; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: celecoxib
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and leucovorin, work in different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. It is not yet known whether fluorouracil and leucovorin are more effective with or without celecoxib in treating resected stage III adenocarcinoma (cancer) of the colon.

PURPOSE: This randomized phase III trial is studying celecoxib, fluorouracil, and leucovorin to see how well they work compared to fluorouracil and leucovorin in treating patients who have undergone surgery for stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare disease-free survival of patients with curatively resected stage III adenocarcinoma of the colon treated with adjuvant fluorouracil and leucovorin calcium with or without celecoxib.

Secondary

* Compare the overall survival, the occurrence of new primary colon cancer, and the development of new polyps in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to ≥ 4 tumor-positive lymph nodes (yes vs no), form of adjuvant chemotherapy (infusional vs bolus), low-dose aspirin for cardiovascular prophylaxis (yes vs no), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fluorouracil and leucovorin calcium IV for up to 6 courses in the absence of disease recurrence or unacceptable toxicity. Patients also receive oral celecoxib twice daily.
* Arm II: Patients receive oral placebo twice daily and fluorouracil and leucovorin calcium as in arm I.

In both arms, treatment with celecoxib or placebo continues for 3 years in the absence of disease recurrence or unacceptable toxicity.

Patients are followed annually for 2 years.

PROJECTED ACCRUAL: A total of 1,450 patients (725 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon

  * 15 cm above anal verge
  * Stage III disease (any pT, N1-2, M0)
* No rectal cancer
* Must have undergone curative radical resection (R0 resection) within the past 6 weeks

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST ≤ 5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* None of the following conditions within the past 6 months:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic congestive heart failure
  * Serious uncontrolled cardiac arrhythmia
  * Cerebrovascular accident or transient ischemic attack
  * Deep vein thrombosis
  * Other significant thromboembolic event

Pulmonary

* No pulmonary embolism within the past 6 months

Gastrointestinal

* No active gastric or duodenal ulceration within the past year
* No gastrointestinal bleeding within the past year
* No partial or complete bowel obstruction
* No known chronic malabsorption
* No active inflammatory bowel disease or chronic diarrhea (more than 4 stools/day)

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No AIDS-related illness
* No prior hypersensitivity to fluorouracil, leucovorin calcium, celecoxib, other COX-2 inhibitors, NSAIDs, salicylates, or sulfonamides
* No other severe acute or chronic medical condition or laboratory abnormality that would preclude study participation, study drug administration, or study results interpretation
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* No concurrent active infection
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent sargramostim (GM-CSF) or molgramostim

Chemotherapy

* Not specified

Endocrine therapy

* No more than 4 weeks of concurrent orally/nasally inhaled steroids over a 6-month period

  * Concurrent mometasone (or fluticasone) allowed if patients require ≥ 4 weeks of inhaled steroid therapy
* At least 30 days since other prior steroids
* No concurrent hormonal therapy

Radiotherapy

* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* No prior total colectomy or other major surgery that would result in substantial alteration in transit to absorption of oral medication

Other

* More than 30 days since prior investigational medication
* No prior systemic anticancer treatment for colon cancer
* No concurrent prophylactic fluconazole
* No concurrent lithium
* No concurrent chronic* use of full dose aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), or cyclo-oxygenase-2 (COX-2) inhibitors

  * Aspirin at cardioprotective doses (i.e., 80 mg daily or equivalent) allowed
* No concurrent participation in any other clinical study
* No other concurrent experimental agents (e.g., other COX-2 inhibitors, matrix metalloproteinase inhibitors, inhibitors of the vascular endothelial growth factor/Flk-1 pathway, or inhibitors of the epidermal growth factor receptor pathway) NOTE: *Chronic use is defined as a frequency of 7 consecutive days (1 week) for more than 3 weeks/year or more than 21 days throughout the year

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-03; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Disease-free survival as measured by Logrank every 3 months in year 1, every 6 months in years 2-3, and annually thereafter

SECONDARY OUTCOMES:
Overall survival as measured by Logrank every 3 months in year 1, every 6 months in years 2-3, and annually thereafter
Time occurrence of new primary colon cancer and new polyps as measured by Logrank every 3 months in year 1, every 6 months in years 2-3, and annually thereafter
Toxicity as measured by CTC AE version 2.0 every 3 months in year 1, every 6 months in years 2-3, and annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J.H. van de Velde, MD, PhD, FRCS, FRCPS, Study Chair — Leiden University Medical Center; Dirk J. Richel, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Michel Ducreux, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (36):
- Austria (7):
  - Karl-Franzens-University Graz, Graz
  - Innsbruck Universitaetsklinik, Innsbruck
  - Krankenhaus der Elisabethinen, Linz
  - St. Vincent's Hospital, Linz Donau
  - Landeskrankenanstalten - Salzburg, Salzburg
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Allgemeines Krankenhaus, Wiener Neustadt
- Belgium (6):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Hopital de Jolimont, Haine-Saint-Paul
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - St. Elizabeth Ziekenhuis, Turnhout
- Netherlands (23):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Gelre Ziekenhuizen - Lokatie Lukas, Apeldoorn
  - Rijnstate Hospital, Arnhem
  - Ziekenhuis Lievensberg, Bergen op Zoom
  - Deventer Ziekenhuisen, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Ziekenhuis St Jansdal, Harderwijk
  - Leiden University Medical Center, Leiden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
  - Waterlandziekenhuis, Purmerend
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Erasmus MC - Sophia Children's Hospital, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Schieland Ziekenhuis, Schiedam
  - Ziekenhuis de Honte, Terneuzen
  - Medisch Centrum Haaglanden, The Hague
  - Streekziekenhuis Koningin Beatrix, Winterswyk
  - Isala Klinieken - locatie Weezenlanden, Zwolle